CLINICAL TRIAL: NCT06871657
Title: Alveolar Ridge Expansion During Indirect Sinus Lift Procedures--A Comparison of Two Surgical Techiques
Brief Title: Comparing Two Surgical Techniques for Building Up the Bone Where a Dental Implant is to Be Placed
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Binnaz Leblebicioglu, Professor, Ohio State University
Other Study IDs: 2023H0106
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Dental Implant; Sinus Floor Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Osseodensification: Patients who are having the sinus lift procedure using the osseodensification technique
  Interventions: Procedure: Sinus lift using osseodensification technique
- Osseocondensation: Patients who are having the sinus lift procedure using the osseocondensation technique
  Interventions: Procedure: Sinus lift using the osseocondensation technique

INTERVENTIONS:
Procedure: Sinus lift using osseodensification technique — Osseodensification dislocates existing bone into trabeculated space by using a bur that turns in anti-clockwise direction. The procedure itself is not part of the research, but is the intervention of interest to the study.
  Groups: Osseodensification
Procedure: Sinus lift using the osseocondensation technique — This procedure is performed by using osteotome hand instruments. The procedure itself is not part of the research, but is the intervention of interest to the study.
  Groups: Osseocondensation

SUMMARY:
The goal of this observational study is to compare two techniques routinely used to increase bone volume in the jaw prior to placing a dental implant, called osseocondensation and osseodensification. The study participants are healthy adults who are planning to get a dental implant. The main questions it aims to answer are:

* Is there a difference in wound closure and soft tissue healing following implant placement using osseocondensation versus osseodensification?
* Is there a difference in bone density around implants placed with osseocondensation versus osseodensification?
* Is there a difference in patient experience during surgery and early phases of healing with osseocondensation versus osseodensification? Researchers will compare implant sites where the osseocondensation technique was used to sites where the osseodensification technique was used to see if there are differences in the outcomes.

It is important to note that the research study will not affect what treatment the participants get. The choice of which technique to use will be made by the dentist who is treating them, based on their clinical judgement. The researchers will only compare the outcomes for the techniques.

For the research study, participants will undergo additional clinical measurements besides those done as the normal post-operative checks, and will fill out questionnaires about their experiences with the procedures. Getting the bone-increasing procedure and getting the dental implant are not part of the research study.

DETAILED DESCRIPTION:
Osseocondensation procedure is a surgical technique developed as an alternative to direct sinus lifting, and it is mainly involved in preparing an implant bed without performing any ostectomy. This is a technique preferred to allow the placement of longer and larger dental implants, especially in posterior upper jaws. The target is to increase the density and the volume of the spongiosa bone at apical-coronal and buccal-lingual dimensions through compression. Although success of this surgical technique has been reported through clinical studies and case reports, some complications such as vertigo have been also documented. Osseodensification technique has been recently developed as an alternative to osseocondensation. This technique uses a special drilling protocol in which the bur turns anti-clockwise and pushes the bone into the trabeculated space instead of using an osteotome. There are several in vitro, in vivo, and clinical studies exploring integrity of bone-implant interface following implant placement through osseodensification technique. However, to the investigators' knowledge, there are no clinical studies comparing this procedure to bone condensation through conventional osteotome technique. Thus, the aim of this study is to compare early healing outcomes of implants placed by using osseocondensation and osseodensification techniques.

Both surgical techniques are currently used interchangeably. The outcomes of these procedures have not been compared within the same study. Thus, the investigators believe that a clinical study comparing these two protocols for early wound healing and bone remodeling would allow clinicians to make evidence-based choices in practice.

Working hypothesis is that there are no patient centered, clinical and radiographic differences between osseocondensation and osseodensification in early peri-implant wound healing outcomes and implant stability. Specific aims: 1. To determine wound closure and soft tissue healing following implant placement by using osseocondensation and osseodensification techniques. 2. To determine changes in CBCT bone density around implant placed with osseocondensation and osseodensification techniques. 3. To evaluate patient centered outcomes during surgery and early phases of wound healing following implant placement with osseocondensation and osseodensification.

Surgical technique being used in this study will be determined by the surgeon as part of standard care (patient and site-specific indications). *Research related procedures: - Radiographic and clinical measurements and recording of the alveolar ridge prior to surgery (dental radiographs and CBCT are routinely obtained as standard of care. The investigators will be using these documents to complete more in-depth analysis of the bone). - Clinical recording of the measurements for the alveolar ridge dimensions after flap elevation and after ridge expansion (this is routinely done as standard of care. The investigators will be recording it for research purpose). - Details of the surgery including bone quality (reported by surgeon), presence of buccal dehiscence/fenestration, the need of additional bone grafting of the ridge, the indications for barrier membrane placement. - Recording of implant stability by recording torque value and/or Osstell value (initial implant stability is an important parameter for the success of the implant and is routinely determined as standard care. The investigators will be recording it as part of the study). - Questions designed to evaluate patient experience (pain and discomfort during and after surgery).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Systemically healthy
* No contraindications for implant placement surgery
* No chronic sinus problems
* Non-smoker
* Minimum ridge width of 3 mm and ridge height of 5 mm

Exclusion Criteria:

* need for ENT specialist clearance due to active problems in relation to ear, not, throat related chronic problems
* sufficient bone volume to perform implant placement without ridge augmentation
* Require guided bone regeneration prior to implant placement
* Need to wear a removable temporary restoration during healing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Graduate Periodontics Clinic at The Ohio State University College of Dentistry who have been treatment-planned for a dental implant and who require an indirect sinus lift procedure prior to implant placement.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in ridge dimensions | Day of surgery and day of uncovery (4-6 months post-surgery)
  Dimensions of the alveolar ridge, determined by measurements on the surgical stent and the CBCT images
Change in Bone Density | Day of procedure and day of uncovery (4-6 months post-operative)
  Bone density around the dental implant, measured via CBCT

SECONDARY OUTCOMES:
Initial Implant Stability | Intraoperative
  Implant stability by measurement of torque value and/or Osstell value, immediately following ridge augmentation and implant placement
Final Implant Stability | 4-6 months post-surgery
  Implant stability by measurement of torque value and/or Osstell value, at implant uncovery appointment 4-6 months post-surgery
Healing Score Index 8-10 days PO | 8-10 days following the surgical procedure
  Pippi modification of Landry wound healing index):
  * presence/absence of redness;
  * presence/absence of granulation tissue;
  * presence/absence of suppuration;
  * presence/absence of swelling;
  * degree of tissue epithelialization (partial/complete);
  * presence/absence of bleeding;
  * presence/absence of pain on palpation.
  * presence/absence of plaque (% of plaque positive surfaces) Performed at first follow-up appointment, 8-10 days post surgery
Healing Score Index 6-8 weeks PO | 6-8 weeks following the surgical procedure
  Pippi modification of Landry wound healing index):
  * presence/absence of redness;
  * presence/absence of granulation tissue;
  * presence/absence of suppuration;
  * presence/absence of swelling;
  * degree of tissue epithelialization (partial/complete);
  * presence/absence of bleeding;
  * presence/absence of pain on palpation.
  * presence/absence of plaque (% of plaque positive surfaces) Performed at second follow-up appointment, 6-8 weeks days post surgery
Wound Healing 8-10 days PO | 8-10 days following the surgical procedure
  Clinical wound healing will be scored as yes or no for each of the following wound healing parameters:
  * Mature wound healing, defined as complete wound closure without other significant findings.
  * Erythema, defined as increased redness compared to adjacent non-operated sites
  * Bleeding, defined as presence of spontaneous bleeding at the wound site
  * Graft mobility, defined as loose subgingival bone graft material evaluated by gentle palpation using a UNC-15 probe {if grafting was done during surgery}
  * Suppuration, defined as presence of pus or discharge at the wound site
  * Necrosis, defined as any visual soft and/or hard tissue necrosis at the wound site
  * Clinical wound exposure( ____ mm)and closure and hydrogen peroxide test(+/-) Assessment performed 8-10 days after surgery
Wound Healing 6-8 weeks PO | 6-8 weeks following the surgical procedure
  Clinical wound healing will be scored as yes or no for each of the following wound healing parameters:
  * Mature wound healing, defined as complete wound closure without other significant findings.
  * Erythema, defined as increased redness compared to adjacent non-operated sites
  * Bleeding, defined as presence of spontaneous bleeding at the wound site
  * Graft mobility, defined as loose subgingival bone graft material evaluated by gentle palpation using a UNC-15 probe {if grafting was done during surgery}
  * Suppuration, defined as presence of pus or discharge at the wound site
  * Necrosis, defined as any visual soft and/or hard tissue necrosis at the wound site
  * Clinical wound exposure( ____ mm)and closure and hydrogen peroxide test(+/-) Assessment performed 6-8 weeks after surgery
Patient Experience Day of Surgery | surgical procedure
  Patient centered evaluation immediately after surgery (if not sedated)
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Any other reported issues
Patient Experience 8-10 Days PO | 8-10 days after surgery
  Patient centered outcomes:
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Swelling (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * The need for analgesics (0=none; 1= first 2 days; 2= first five days; 3= more than five days)
  * Any reported issues
  Evaluated at first post-operative visit, 8-10 days following the surgical procedure
Patient Experience 6-8 Weeks PO | 6-8 weeks after surgery
  Patient centered outcomes:
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Swelling (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * The need for analgesics (0=none; 1= first 2 days; 2= first five days; 3= more than five days)
  * Any reported issues
  Evaluated at second post-operative visit
Patient Experience 4-6 months PO | 4-6 months after surgery
  Patient centered outcomes:
  * Discomfort level (0 = no; 1 = mild; 2 = moderate; 3 = severe)
  * Pain (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * Swelling (0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  * The need for analgesics (0=none; 1= first 2 days; 2= first five days; 3= more than five days)
  * Any reported issues
  Evaluated at implant uncovery appointment

CONTACTS AND LOCATIONS:
Overall Officials: Binnaz Leblebicioglu, DDS, MS, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Dentistry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No